CLINICAL TRIAL: NCT01344447
Title: Multicenter, Open-label Study to Evaluate the Safety and Efficacy (by Blinded Reading) of Contrast-Enhanced Magnetic Resonance Angiography (MRA) After a Single Intravenous Injection of 0.1 mmol/kg Gadobutrol in Subjects With Known or Suspected Vascular Disease of the Supra-aortic Vessels
Brief Title: Gadobutrol Enhanced MRA of the Supra-aortic Vessels
Acronym: GEMSAV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14607; 2010-023001-36 (EudraCT Number)
Record Dates: First submitted 2011-04-05; First posted 2011-04-29 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Carotid Stenosis
Keywords: Supra-aortic vascular disease; MRA; CTA; Males and females aged 18 years or older; Stroke; Transient Ischemic Attack (TIA)
MeSH Terms: conditions — Carotid Stenosis; Stroke; Ischemic Attack, Transient | interventions — gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Gadobutrol (Gadovist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadovist, BAY86-4875) — A single bolus injection of approx. 0.1mmol/kg

SUMMARY:
Subjects referred for a routine CTA (computed tomography angiography) or MRA (magnetic resonance angiography) will be invited to participate in the study and subjects will be involved in the study for between 2 and 12 days. Two to three visits to the study doctor will be required.

This study will compare the diagnostic results of Gadobutrol enhanced MRA images with MRA images taken without contrast agent using images from a CTA as the standard of reference, which may have been performed up to 60 days prior to enrolment. If a CTA has not been performed in this prior time period, a CTA is required for the study.

MRA and CTA images will be collected for an independent review (blinded read).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 18 years and older
* Any of the following:

  * Known or suspected supra-aortic arterial disease based on:

    * Prior stroke
    * Transient ischemic attack (TIA)
    * Amaurosis Fugax (transient monocular blindness)
  * Referred for evaluation of any supra-aortic vessel (for clinically significant stenosis)
  * Follow-up for a stent in a supra-aortic vessel
  * Prior imaging study (CTA or ultrasound) showing ≥ 50% stenosis of a supra-aortic vessel segment (within 60 days before consent). The proportion of subjects with positive disease (determined by the investigator, based on CTA or ultrasound) will be monitored during the study, and enrolment may be further restricted to require ≥ 70% stenosis to ensure that overall there are an adequate number of subjects with clinically significant disease for the evaluation of study endpoints.
* Willingness to undergo the routine Contrast Enhanced Magnetic Resonance Angiography [CE MRA] examination with gadobutrol
* Willingness and ability to follow directions and complete all study procedures specified in the protocol
* Females of childbearing potential only: Negative pregnancy test on the day of the MRA before the administration of study drug

Exclusion Criteria:

* Pregnant or nursing (including pumping for storage and feeding)
* Received any other investigational product or participation in any other clinical trial within 30 days before enrollment into this study
* Previous enrollment into this study or into any other Bayer sponsored study using gadobutrol
* Contraindication to the MRA examinations (e.g. inability to hold breath; severe arrhythmias; very low cardiac output, severe claustrophobia, defibrillators or other metallic devices not approved for MRI)
* Contraindication to the use of Gd-containing contrast agents (including subjects with suspicion for or known to have Nephrogenic Systemic Fibrosis [NSF])
* History of severe allergic or anaphylactoid reaction to any allergen including drugs and contrast agents
* Received any contrast agent within 72 hours before the study MRA, or scheduled receipt of any contrast agent within 24 hours after the study MRA (Note: This applies also to a CTA potentially scheduled during the course of the study.)
* Estimated glomerular filtration rate (eGFR) value < 30 ml/min/1.73 m2 derived from a serum creatinine result within 2 weeks before the gadobutrol injection. Any subject on hemodialysis or peritoneal dialysis is excluded from participation. Use the value obtained prior to and closest to the time of the MRA, if there are multiple creatinine values. (Do not use the core lab value if not available prior to the MRA.)
* Acute renal insufficiency of any intensity, either due to hepato-renal syndrome or occurring in the peri-operative liver transplantation period
* Severe cardiovascular disease (e.g. acute myocardial infarction [< 14 days], unstable angina, congestive heart failure New York Heart Association class IV) or known long QT syndrome
* Suspected clinical instability or unpredictability of the clinical course during the study period (e.g. due to previous surgery)
* Scheduled or potentially expected for the period between the CTA and gadobutrol MRA:

  * Any procedure that may alter the MRA or CTA interpretation, or
  * Any interventional or surgical procedure involving the supra-aortic vessels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2011-05-12 (Actual); Primary Completion 2014-05-28 (Actual); Study Completion 2014-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (51):
- United States (15):
  - Tucson, Arizona
  - Jacksonville, Florida
  - Savannah, Georgia
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Jackson, Mississippi
  - Rochester, New York
  - The Bronx, New York
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Memphis, Tennessee
  - Seattle, Washington
  - Madison, Wisconsin
- Argentina (2):
  - Adrogué, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
- Australia (3):
  - New Lambton Heights, New South Wales
  - Clayton, Victoria
  - Parkville, Victoria
- Austria (2):
  - Innsbruck, Tyrol
  - Vienna
- Shanghai, China
- Brno, Czechia
- France (4):
  - Brest
  - Bron
  - Marseille
  - Paris
- Germany (5):
  - Karlsruhe, Baden-Wurttemberg
  - Augsburg, Bavaria
  - Erlangen, Bavaria
  - Münster, North Rhine-Westphalia
  - Jena, Thuringia
- Italy (6):
  - Aosta, Aosta Valley
  - Ferrara, Emilia-Romagna
  - Rome, Lazio
  - Catania, Sicily
  - Massa-Carrara, Tuscany
  - Venezia, Veneto
- Poland (4):
  - Bydgoszcz
  - Lodz
  - Warsaw
  - Wroclaw
- South Korea (2):
  - Donggu, Gwangju Gwang''yeogsi
  - Seoul
- Sweden (2):
  - Linköping
  - Uppsala
- Sankt Gallen, Canton of St. Gallen, Switzerland
- Turkey (Türkiye) (3):
  - Antalya
  - Erzurum
  - Istanbul

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 56 study centers in 14 countries, between 12 May 2011 (first participant first visit) and 28 May 2014 (last participant last visit).
Pre-assignment Details: Of 504 participants screened, 17 did not complete screening; due to screen failure in 6, consent withdrawal in 6 and other reasons in 5 participants. Of 487 participants assigned to treatment, 479 received study drug and 8 prematurely terminated due to adverse event in 7 participants, and other reason in 1 participant.
Groups:
- Gadobutrol (Gadavist, BAY 86-4875): Gadobutrol was administered to all participants receiving study drug at the standard dose of 0.1 millimole per kilogram (mmol/kg) body weight (BW) by single intravenous (IV) bolus injection. During the course of the study, non-contrast MRA images were obtained before the administration of gadobutrol, and gadobutrol-enhanced MRA images were obtained after injection.
Period: Overall Study
Arm/Group | Gadobutrol (Gadavist, BAY 86-4875)
Started | 479 (Participant received study drug; Safety analysis set)
Fulfilled Requirement of FAS Population | 457 (Full Analysis Set (FAS))
Completed | 471
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — The contrast was not seen | 1
Not completed — Physician Decision | 1
Not completed — MRA unsuccessful | 1
Not completed — Bolus tracking failed | 1
Not completed — Error of power injector | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gadobutrol (Gadavist, BAY 86-4875)
Number analyzed (Participants) | 479
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (10)
Age, Customized [Number; unit: participants]
  <45 years | 9
  45-64 years | 155
  >=65 years | 315
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167
  Male | 312
Baseline Weight [Mean (Standard Deviation); unit: kilogram] | 76.0 (14.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Assessable Vascular Segments Using Gadobutrol-Enhanced MRA and Unenhanced MRA
Description: Each vascular segment was visualized using unenhanced MRA and gadobutrol-enhanced MRA, characterized by the on-site investigators, three independent blinded readers (BR) (BR 1, BR 2 and BR 3) and majority readers (the outcome determined by at least two of the blinded readers). A segment was assessable if it was visualized along its entire length and if any region of stenosis, was measured reliably. There were 21 segments of the supra-aortic arteries assessed per participant.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS
Measure: Number; unit: percentage of segments
Units Other Than Participants: segments
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 457 | 457
Number analyzed (segments) | 9597 | 9597
percentage of segments
  Majority reader | 95.0 | 72.7
  Blinded reader 1 | 88.2 | 24.4
  Blinded reader 2 | 94.9 | 75.3
  Blinded reader 3 | 97.4 | 82.4
  Clinical investigators | 97.0 | 78.6
Statistical Analysis 1: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Majority reader; Superiority analysis; The percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Superiority or Other; p < 0.0001, McNemar; Cluster adjusted McNemar; Percentage difference = 22.3, 95.1% CI 2-sided [lower limit 20.4] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 2: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Blinded reader 1; Superiority analysis; The percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Superiority or Other; p < 0.0001, McNemar; Cluster adjusted McNemar; Percentage difference = 63.8, 95.1% CI 2-sided [lower limit 60.9] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 3: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Blinded reader 2; Superiority analysis; The percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Superiority or Other; p < 0.0001, McNemar; Cluster adjusted McNemar; Percentage difference = 19.6, 95.1% CI 2-sided [lower limit 17.8] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 4: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Blinded reader 3; Superiority analysis; The percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Superiority or Other; p < 0.0001, McNemar; Cluster adjusted McNemar; Percentage difference = 15.0, 95.1% CI 2-sided [lower limit 13.3] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 5: Comparison: Gadobutrol-enhanced MRA vs Unenhanced MRA; Clinical investigator; Superiority analysis; The percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Superiority or Other; p < 0.0001, McNemar; Cluster adjusted McNemar; Percentage difference = 18.5, 95.1% CI 2-sided [lower limit 16.5] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)

2. Primary Outcome: Sensitivity for Detection of Clinically Significant Disease Using Gadobutrol-Enhanced MRA and Unenhanced MRA
Description: Clinically significant disease was defined as 70 to 99% stenosis of a segment, but not occluded, as assessed by the standard of reference (SoR) (computed tomographic angiography [CTA]; blinded readers). This was determined using the North American Symptomatic Carotid Endarterectomy Trial (NASCET) criteria. For each segment, the most severe stenosis/narrowing was identified and considered for the evaluation of clinically significant disease. In case of multiple stenosis in any one segment, the most severe stenosis in the segment was recorded.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS; in below table, "n/n" signifies the number of participants/segments that were evaluable in specified category of each group.
Measure: Number; unit: percentage of sensitivity
Units Other Than Participants: segments
Arm/Group | Gadobutrol-enhanced MRA | Non-contrast MRA
Number analyzed (Participants) | 238 | 238
Number analyzed (segments) | 297 | 297
percentage of sensitivity
  Majority reader (n=141/158) | 60.1 | 54.4
  Blinded reader 1 (n=141/158) | 59.5 | 54.4
  Blinded reader 2 (n=141/158) | 59.5 | 54.1
  Blinded reader 3 (n=141/158) | 58.2 | 55.7
  Clinical investigators (n=238/297) | 60.9 | 39.4
Statistical Analysis 1: Comparison: Gadobutrol-enhanced MRA vs Non-contrast MRA; Majority reader; The percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 5.7, 95.1% CI 2-sided [lower limit -3.6] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 2: Comparison: Gadobutrol-enhanced MRA vs Non-contrast MRA; Blinded reader 1; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 5.1, 95.1% CI 2-sided [lower limit -5.4] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 3: Comparison: Gadobutrol-enhanced MRA vs Non-contrast MRA; Blinded reader 2; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 5.1, 95.1% CI 2-sided [lower limit -4.7] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 4: Comparison: Gadobutrol-enhanced MRA vs Non-contrast MRA; Blinded reader 3; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 3.2, 95.1% CI 2-sided [lower limit -5.9] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 5: Comparison: Gadobutrol-enhanced MRA vs Non-contrast MRA; Clinical investigator; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 21.5, 95.1% CI 2-sided [lower limit 14.1] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)

3. Primary Outcome: Specificity for Exclusion of Clinically Significant Disease Using Gadobutrol-Enhanced MRA and Unenhanced MRA
Description: Clinically significant disease was defined as 70 to 99% stenosis of a segment, but not occluded, as assessed by the SoR (CTA; blinded readers). This was determined using the NASCET criteria. For each segment, the most severe stenosis/narrowing was identified and considered for the evaluation of clinically significant disease. In case of multiple stenosis in any one segment, the most severe stenosis in the segment was recorded.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS; in below table, "n/n" signifies the number of participants/segments that were evaluable in specified category of each group if it varies from "Number of participants/segments analyzed".
Measure: Number; unit: percentage of specificity
Units Other Than Participants: segments
Arm/Group | Gadobutrol-enhanced MRA | Non-contrast MRA
Number analyzed (Participants) | 457 | 457
Number analyzed (segments) | 9321 | 9321
percentage of specificity
  Majority reader (n=457/9321) | 96.1 | 87.3
  Blinded reader 1 (n=457/9321) | 92.0 | 61.7
  Blinded reader 2 (n=457/9321) | 94.7 | 85.1
  Blinded reader 3 (n=457/9321) | 96.7 | 89.1
  Clinical investigators (n=457/9133) | 98.1 | 89.1
Statistical Analysis 1: Comparison: Gadobutrol-enhanced MRA vs Non-contrast MRA; Majority reader; The percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 8.8, 95.1% CI 2-sided [lower limit 7.7] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 2: Comparison: Gadobutrol-enhanced MRA vs Non-contrast MRA; Blinded reader 1; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 30.3, 95.1% CI 2-sided [lower limit 28.6] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 3: Comparison: Gadobutrol-enhanced MRA vs Non-contrast MRA; Blinded reader 2; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 9.7, 95.1% CI 2-sided [lower limit 8.5] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 4: Comparison: Gadobutrol-enhanced MRA vs Non-contrast MRA; Blinded reader 3; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 7.6, 95.1% CI 2-sided [lower limit 6.6] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)
Statistical Analysis 5: Comparison: Gadobutrol-enhanced MRA vs Non-contrast MRA; Clinical investigator; the percentage difference was calculated as gadobutrol-enhanced minus unenhanced MRA; Test type: Non-Inferiority or Equivalence — using a -7.5% non-inferiority margin; The cluster-adjusted two-sided 95% CI; Percentage difference = 9.1, 95.1% CI 2-sided [lower limit 7.9] (Not Appropriate, upper intervals were not used in the statistical analysis and were not of interest for the study.)

4. Primary Outcome: Minimum Gadobutrol Performance for Sensitivity: Sensitivity > 50%
Description: Clinically significant disease was defined as 70 to 99% stenosis of a segment, but not occluded as assessed by the SoR (CTA; blinded readers). For each segment, the most severe stenosis/narrowing was identified and considered for the evaluation of clinically significant disease. Gadobutrol minimum performance criteria was based on a stenosis of 50% calculated from the native vessel diameter.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS; in below table, "n/n" signifies the number of participants/segments that were evaluable in specified category.
Measure: Number; unit: percentage of sensitivity
Units Other Than Participants: segments
Arm/Group | Gadobutrol-enhanced MRA
Number analyzed (Participants) | 230
Number analyzed (segments) | 283
percentage of sensitivity
  Majority reader (n=135/149) | 61.7
  Blinded reader 1 (n=132/146) | 60.3
  Blinded reader 2 (n=139/156) | 59.6
  Blinded reader 3 (n=140/155) | 58.7
  Clinical investigators (n=230/283) | 61.5
Statistical Analysis 1: Comparison: Gadobutrol-enhanced MRA; Majority reader; Test type: Superiority or Other; One sided 95.1% confidence interval; percentage = 61.7, 95.1% CI 1-sided [lower limit 55.3]
Statistical Analysis 2: Comparison: Gadobutrol-enhanced MRA; Blinded Reader 1; Test type: Superiority or Other; One sided 95.1% confidence interval; percentage = 60.3, 95.1% CI 1-sided [lower limit 53.6]
Statistical Analysis 3: Comparison: Gadobutrol-enhanced MRA; Blinded Reader 2; Test type: Superiority or Other; One sided 95.1% confidence interval; percentage = 59.6, 95.1% CI 1-sided [lower limit 53.1]
Statistical Analysis 4: Comparison: Gadobutrol-enhanced MRA; Blinded Reader 3; Test type: Superiority or Other; One sided 95.1% confidence interval; percentage = 58.7, 95.1% CI 1-sided [lower limit 52.2]
Statistical Analysis 5: Comparison: Gadobutrol-enhanced MRA; Clinical investigator; Test type: Superiority or Other; One sided 95.1% confidence interval; percentage = 61.5, 95.1% CI 1-sided [lower limit 56.7]

5. Primary Outcome: Minimum Gadobutrol Performance for Specificity: Specificity > 50%
Description: as for outcome 4
Time Frame: Images were taken pre-injection and post-injection
Population: FAS; in below table, "n/n" signifies the number of participants/segments that were evaluable in specified category.
Measure: Number; unit: percentage of specificity
Units Other Than Participants: segments
Arm/Group | Gadobutrol-enhanced MRA
Number analyzed (Participants) | 457
Number analyzed (segments) | 8926
percentage of specificity
  Majority reader (n=457/8805) | 98.0
  Blinded reader 1 (n=444/8225) | 97.6
  Blinded reader 2 (n=457/8844) | 97.2
  Blinded reader 3 (n=457/9079) | 98.0
  Clinical investigators (n=457/8926) | 99.2
Statistical Analysis 1: Comparison: Gadobutrol-enhanced MRA; Majority reader; Test type: Superiority or Other; One sided 95.1% confidence interval; percentage = 98.0, 95.1% CI 1-sided [lower limit 97.7]
Statistical Analysis 2: Comparison: Gadobutrol-enhanced MRA; Blinded Reader 1; Test type: Superiority or Other; One sided 95.1% confidence interval; percentage = 97.6, 95.1% CI 1-sided [lower limit 97.3]
Statistical Analysis 3: Comparison: Gadobutrol-enhanced MRA; Blinded Reader 2; Test type: Superiority or Other; One sided 95.1% confidence interval; percentage = 97.2, 95.1% CI 1-sided [lower limit 96.9]
Statistical Analysis 4: Comparison: Gadobutrol-enhanced MRA; Blinded Reader 3; Test type: Superiority or Other; One sided 95.1% confidence interval; percentage = 98.0, 95.1% CI 1-sided [lower limit 97.7]
Statistical Analysis 5: Comparison: Gadobutrol-enhanced MRA; Clinical investigator; Test type: Superiority or Other; One sided 95.1% confidence interval; percentage = 99.2, 95.1% CI 1-sided [lower limit 98.9]

6. Secondary Outcome: Vessel Diameter (Millimeter [mm]) at the Normal Point and the Narrowest Point in Gadobutrol-Enhanced MRA, Unenhanced MRA and CTA Images
Description: The segment reduction in diameter (DIA) of greater than 10% was considered abnormal and measured. The diameter of each of these abnormal segments was measured using electronic calipers (perpendicular to the long axis of the vessel) at the point of most severe stenosis within each segment. Mean of vessel diameters was calculated by segment separately for CTA and MRA readers. For ease of expression, the following abbreviations will be used: Diameter (DIA), Blinded Reader (BR), Clinical Investigator (CI).
Time Frame: Images were taken pre-injection and post-injection
Population: FAS; Number of participants/segments analyzed in below ordered categories (Normal-BRs; Narrowest-BRs; Normal-CIs; Narrowest-CIs) in Enhanced MRA group was 457/6182, 457/6182, 419/1361, 419/1352 respectively; in Unenhanced MRA group was 455/4776, 455/4776, 367/989, 367/980 respectively; in CTA was 442/3158, 442/3158, 419/1569, 419/1555 respectively.
Measure: Mean (Standard Deviation); unit: millimeter(s) (mm)
Arm/Group | Gadobutrol-Enhanced MRA | Unenhanced MRA | Computed Tomographic Angiography
Number analyzed (Participants) | 457 | 455 | 442
millimeter(s) (mm)
  Vessel DIA at normal point: BRs | 4.88 (1.90) | 4.33 (1.53) | 4.98 (2.08)
  Vessel DIA at narrowest point: BRs | 3.23 (1.54) | 2.66 (1.34) | 3.00 (1.50)
  Vessel DIA at normal point: CIs | 4.81 (1.78) | 4.54 (1.58) | 5.17 (2.02)
  Vessel DIA at narrowest point: CIs | 2.42 (1.37) | 2.31 (1.21) | 2.68 (1.62)
Statistical Analysis 1: Comparison: Unenhanced MRA vs Computed Tomographic Angiography; CTA Minus Unenhanced MRA for blinded Reader on vessel DIA at normal point; Test type: Superiority or Other; Mean Difference; Diameter difference = 0.21, Standard Deviation 0.80
Statistical Analysis 2: Comparison: Gadobutrol-Enhanced MRA vs Computed Tomographic Angiography; CTA minus Gadobutrol-Enhanced MRA for blinded reader on vessel DIA at normal point; Test type: Superiority or Other; Mean Difference; Diameter difference = 0.00, Standard Deviation 0.79
Statistical Analysis 3: Comparison: Unenhanced MRA vs Computed Tomographic Angiography; CTA minus Unenhanced MRA for blinded reader on vessel DIA at narrowest point; Test type: Superiority or Other; Mean Difference; Diameter difference = 0.29, Standard Deviation 0.87
Statistical Analysis 4: Comparison: Gadobutrol-Enhanced MRA vs Computed Tomographic Angiography; CTA minus Gadobutrol-Enhanced MRA for blinded reader on vessel DIA at narrowest point; Test type: Superiority or Other; Mean Difference; Diameter difference = 0.01, Standard Deviation 0.80
Statistical Analysis 5: Comparison: Unenhanced MRA vs Computed Tomographic Angiography; CTA minus Unenhanced MRA for clinical investigators on vessel DIA at normal point; Test type: Superiority or Other; Mean Difference; Diameter difference = 0.48, Standard Deviation 0.98
Statistical Analysis 6: Comparison: Gadobutrol-Enhanced MRA vs Computed Tomographic Angiography; CTA minus Gadobutrol-enhanced MRA for clinical investigators on vessel DIA at normal point; Test type: Superiority or Other; Mean Difference; Diameter difference = 0.33, Standard Deviation 1.01
Statistical Analysis 7: Comparison: Unenhanced MRA vs Computed Tomographic Angiography; CTA minus Unenhanced MRA for clinical investigators on vessel DIA at narrowest point; Test type: Superiority or Other; Mean Difference; Diameter difference = 0.02, Standard Deviation 0.81
Statistical Analysis 8: Comparison: Gadobutrol-Enhanced MRA vs Computed Tomographic Angiography; CTA minus Gadobutrol-enhanced MRA for clinical investigators on vessel DIA at narrowest point; Test type: Superiority or Other; Mean Difference; Diameter difference = 0.11, Standard Deviation 0.79

7. Secondary Outcome: The Percentage of Segments With Artifacts Presence
Description: Artifacts were collected for the MRA images on a segmental basis.
Time Frame: Images were taken pre-injection and post-injection
Population: Evaluable participants in FAS
Measure: Number; unit: percentage of segments
Units Other Than Participants: segments
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 457 | 457
Number analyzed (segments) | 9821 | 9552
percentage of segments
  Blinded reader 1 | 46.6 | 97.1
  Blinded reader 2 | 14.0 | 54.9
  Blinded reader 3 | 16.2 | 41.2

8. Secondary Outcome: Types of Artifacts on a Segment Basis by Blinded Reader 1
Description: The following types of artifacts were considered: Motion artifact (including pulsatility, breathing, swallowing), venous opacification, saturation artifact (for example [eg], in-plane flow, turbulence, dephasing, saturation band), susceptibility artifacts (including devices, eg, stents), ringing artifact (eg, bands), bolus timing error, and other (artifact not specified above or no artifact).
Time Frame: Images were taken pre-injection and post-injection
Population: Participants in FAS with artifacts presence.
Measure: Number; unit: percentage of segments
Units Other Than Participants: segments
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 457 | 457
Number analyzed (segments) | 9821 | 9552
percentage of segments
  Motion artifact | 18.6 | 41.9
  Venous opacification | 9.8 | 0.8
  Saturation artifact | 21.6 | 38.2
  Susceptibility artifacts | 0.1 | 0.2
  Ringing artifact | 0.5 | 29.3
  Bolus timing error | 4.3 | 4.0
  Other | 9.3 | 48.0

9. Secondary Outcome: Types of Artifacts on a Segment Basis by Blinded Reader 2
Description: as for outcome 8
Time Frame: Images were taken pre-injection and post-injection
Population: Participants in FAS with artifacts presence.
Measure: Number; unit: percentage of segments
Units Other Than Participants: segments
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 457 | 457
Number analyzed (segments) | 9821 | 9552
percentage of segments
  Motion artifact | 5.6 | 39.8
  Venous opacification | 5.7 | 0.3
  Saturation artifact | 2.0 | 24.5
  Susceptibility artifacts | 0.8 | 3.7
  Ringing artifact | 0.2 | 0.0
  Bolus timing error | 1.1 | 0.0
  Other | 0.5 | 0.3

10. Secondary Outcome: Types of Artifacts on a Segment Basis by Blinded Reader 3
Description: as for outcome 8
Time Frame: Images were taken pre-injection and post-injection
Population: Participants in FAS with artifacts presence.
Measure: Number; unit: percentage of segments
Units Other Than Participants: segments
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 457 | 457
Number analyzed (segments) | 9821 | 9552
percentage of segments
  Motion artifact | 0.6 | 13.2
  Venous opacification | 1.7 | 0.1
  Saturation artifact | 13.8 | 39.4
  Susceptibility artifacts | 0.2 | 0.5
  Ringing artifact | 0.6 | 6.4
  Bolus timing error | 1.6 | 0.4
  Other | 0.4 | 0.1

11. Secondary Outcome: The Percentage of Location of Stenosis (>=70%) in the Proximal Segments Assessed by Gadobutrol-Enhanced MRA and Unenhanced MRA
Description: Location within a segment was based on the point of greatest stenosis and was recorded for stenosis >=70% (including occlusions) as: - At the bifurcation or proximal origin of a segment (occlusion proximal to the origin of the segment); - Within 5 mm of the bifurcation or proximal origin of a segment; - Beyond 5 mm from the bifurcation or proximal origin of a segment.
Time Frame: Images were taken pre-injection and post-injection
Population: Evaluable participants in FAS; in the below table, "n" signifies number of locations that were evaluable for the specified category of each group.
Measure: Number; unit: pecentage of location
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 457 | 457
pecentage of location
  At the bifurcation: BR 1 (n=353; 89) | 50.4 | 59.6
  At the bifurcation: BR 2 (n=429; 429) | 52.2 | 58.7
  At the bifurcation: BR 3 (n=525; 559) | 44.0 | 54.2
  Within 5 mm of the bifurcation: BR 1 (n=353; 89) | 16.7 | 12.4
  Within 5 mm of the bifurcation: BR 2 (n=429; 429) | 14.7 | 10.7
  Within 5 mm of the bifurcation: BR 3 (n=525; 559) | 34.7 | 27.0
  Beyond 5 mm of the bifurcation: BR 1 (n=353; 89) | 32.9 | 28.1
  Beyond 5 mm of the bifurcation: BR 2 (n=429; 429) | 33.1 | 30.5
  Beyond 5 mm of the bifurcation: BR 3 (n=525; 559) | 21.3 | 18.8

12. Secondary Outcome: Length of Stenosis (>=70%) in the Proximal Segments Assessed by Gadobutrol-Enhanced MRA and Unenhanced MRA
Description: The length of stenosis was based on the most proximal (first point) in a segment where a stenosis exceeded 10% and the most distal point (last point) in the segment where a stenosis exceeded 10%. If a stenosis spanned more than one segment then the measurement was only included to the beginning or end (boundary) of the segment being evaluated. If there was no stenosis of >=70% in a segment then the length was designated as 0.
Time Frame: Images were taken pre-injection and post-injection
Population: Evaluable participants in FAS; this outcome measure was analyzed on a segment basis, in the below table, "n" signifies number of segments that were evaluable for the specified category of each group.
Measure: Mean (Standard Deviation); unit: millimeter(s)
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 457 | 457
millimeter(s)
  Reader 1 (n=290; 66) | 11.26 (11.77) | 13.36 (11.47)
  Reader 2 (n=315; 281) | 6.25 (6.99) | 7.18 (6.07)
  Reader 3 (n=277; 268) | 4.89 (4.69) | 5.36 (3.76)

13. Secondary Outcome: The Percentage of Presence of Secondary Radiologic Indicators for Diagnosis of Clinically Relevant Disease
Description: Each segment was assessed for secondary signs of stenosis for diagnosis of clinically significant disease. The following indicators were considered for the MRA studies: - post-stenotic dilation or ulceration (segmental), - post-stenotic signal dropout, narrowing and intensity reduction, and - thrombus. Each of the three parameters were assessed as present or absent in the region distal to the stenosis. If they were found in any segment distal to the stenosis then they were assessed as present.
Time Frame: Images were taken pre-injection and post-injection
Population: Evaluable participants in FAS; this outcome measure was analyzed on a segment basis, in below table, "n" signifies segments that were evaluable for the specified category of each group.
Measure: Number; unit: percentage of radiologic indicator
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 457 | 457
percentage of radiologic indicator
  Reader 1 (n=9336; 9203) | 3.9 (11.77) | 0.7 (11.47)
  Reader 2 (n=9444; 9177) | 2.8 (6.99) | 2.0 (6.07)
  Reader 3 (n=9285; 9009) | 2.4 (4.69) | 2.7 (3.76)

14. Secondary Outcome: Type of Secondary Radiologic Indicators for Diagnosis of Clinically Relevant Disease
Description: Each segment was assessed for secondary signs of stenosis for diagnosis of clinically significant disease. The following indicators were considered for the MRA studies: - post-stenotic dilation or ulceration (segmental), - post-stenotic signal dropout, narrowing and intensity reduction, and - thrombus. Each of the three parameters were assessed as present or absent in the region distal to the stenosis. If they were found in any segment distal to the stenosis then they were assessed as present. If there were tandem (serial) stenosis in a vessel then the secondary signs were assigned to the stenosis of >=70% that was proximal and closest in proximity to the secondary sign.
Time Frame: Images were taken pre-injection and post-injection
Population: Evaluable participants in FAS; this outcome measure was analyzed on a segment basis, in below table, "n" signifies number of segments with presence of secondary radiologic indicators for the specified category of each group.
Measure: Number; unit: percentage of segments
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 457 | 457
percentage of segments
  Post-stenotic dilation: BR 1 (n=390; 63) | 49.7 (11.77) | 20.6 (11.47)
  Post-stenotic dilation: BR 2 (n=271; 188) | 74.2 (6.99) | 56.4 (6.07)
  Post-stenotic dilation: BR 3 (n=236; 246) | 7.2 (4.69) | 1.6 (3.76)
  Post-stenotic signal dropout: BR 1 (n=390; 63) | 49.5 | 77.8
  Post-stenotic signal dropout: BR 2 (n=271; 188) | 25.5 | 43.6
  Post-stenotic signal dropout: BR 3(n=236; 246) | 92.8 | 98.4
  Thrombus: BR 1 (n=390; 63) | 0.8 | 1.6
  Thrombus: BR 2 (n=271; 188) | 0.4 | 0.0
  Thrombus: BR 3 (n=236; 246) | 0.0 | 0.0

15. Secondary Outcome: Diagnostic Confidence by the Blinded Readers Using Gadobutrol-Enhanced MRA and Unenhanced MRA
Description: Diagnostic confidence was evaluated to determine the level of certainty that the blinded readers assigned to a diagnosis for each segment. This was defined as the degree of confidence that the information on the MRA images represented the true and complete clinical picture of a particular segment. The degree of confidence was rated on a 4-point scale: 1 = Not confident, 2 = Somewhat confident, 3 = Confident, and 4 = Very confident.
Time Frame: Images were taken pre-injection and post-injection
Population: Evaluable participants in FAS; this outcome measure was analyzed on a segment basis, in below table, "n" signifies number of segments that were evaluable for the specified category of each group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 457 | 456
units on a scale
  Reader 1 (n=9408; 9231) | 3.2 (1.0) | 1.3 (0.6)
  Reader 2 (n=9535; 9301) | 2.9 (0.6) | 2.2 (0.9)
  Reader 3 (n=9539; 9302) | 2.8 (0.5) | 2.4 (0.8)

16. Secondary Outcome: The Percentage of Participants With Additional Imaging Studies Recommended by the Blinded Readers and the Clinical Investigator After Evaluation of the Unenhanced and Gadobutrol-Enhanced MRA Images
Description: A measure of diagnostic value was the reduction in the number of additional diagnostic imaging studies recommended/ordered. The clinical investigators and the blinded readers were asked if they would have recommended an additional imaging study for each participant and was recorded.
Time Frame: Images were taken pre-injection and post-injection
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 457 | 457
percentage of participants
  Reader 1 | 71.1 (11.77) | 100.0 (11.47)
  Reader 2 | 44.2 (6.99) | 98.2 (6.07)
  Reader 3 | 22.1 (4.69) | 83.2 (3.76)
  Clinical investigators | 11.2 | 43.1

17. Secondary Outcome: Types of Additional Imaging Studies Recommended by the Blinded Readers After Evaluation of the Unenhanced and Gadobutrol-Enhanced MRA Images - Blinded Reader 1
Description: An additional imaging study recommended was specified from the following list: Non-contrast MRA, Contrast-enhanced MRA, CTA, Ultrasound, Digital subtraction catheter angiogram (DSCA), and Nuclear medicine study.
Time Frame: Images were taken pre-injection and post-injection
Population: Participants in FAS who were recommended for additional imaging studies.
Measure: Number; unit: participants
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 325 | 457
participants
  Non-contrast MRA | 0 (11.77) | 0 (11.47)
  Contrast-enhanced MRA | 64 (6.99) | 448 (6.07)
  CTA | 124 (4.69) | 4 (3.76)
  Ultrasound | 0 | 0
  DSCA | 137 | 5
  Nuclear medicine study | 0 | 0

18. Secondary Outcome: Types of Additional Imaging Studies Recommended by the Blinded Readers After Evaluation of the Unenhanced and Gadobutrol-Enhanced MRA Images - Blinded Reader 2
Description: as for outcome 17
Time Frame: Images were taken pre-injection and post-injection
Population: Participants in FAS who were recommended for additional imaging studies.
Measure: Number; unit: participants
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 202 | 449
participants
  Non-contrast MRA | 50 (11.77) | 2 (11.47)
  Contrast-enhanced MRA | 30 (6.99) | 415 (6.07)
  CTA | 113 (4.69) | 30 (3.76)
  Ultrasound | 0 | 0
  DSCA | 9 | 2
  Nuclear medicine study | 0 | 0

19. Secondary Outcome: Types of Additional Imaging Studies Recommended by the Blinded Readers After Evaluation of the Unenhanced and Gadobutrol-Enhanced MRA Images - Blinded Reader 3
Description: as for outcome 17
Time Frame: Images were taken pre-injection and post-injection
Population: Participants in FAS who were recommended for additional imaging studies.
Measure: Number; unit: participants
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 101 | 380
participants
  Non-contrast MRA | 0 (11.77) | 0 (11.47)
  Contrast-enhanced MRA | 12 (6.99) | 64 (6.07)
  CTA | 88 (4.69) | 316 (3.76)
  Ultrasound | 0 | 0
  DSCA | 1 | 0
  Nuclear medicine study | 0 | 0

20. Secondary Outcome: Types of Additional Imaging Studies Recommended by the Clinical Investigator After Evaluation of the Unenhanced and Gadobutrol-Enhanced MRA Images
Description: as for outcome 17
Time Frame: Images were taken pre-injection and post-injection
Population: Participants in FAS who were recommended for additional imaging studies.
Measure: Number; unit: participants
Arm/Group | Gadobutrol-enhanced MRA | Unenhanced MRA
Number analyzed (Participants) | 51 | 197
participants
  Non-contrast MRA | 1 (11.77) | 0 (11.47)
  Contrast-enhanced MRA | 0 (6.99) | 142 (6.07)
  CTA | 44 (4.69) | 51 (3.76)
  Ultrasound | 1 | 0
  DSCA | 5 | 4
  Nuclear medicine study | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time the consent was signed until 24 (+/-6) hours follow-up after the study MRA but was continued until completion of the CTA in those participants who had the CTA performed after the MRA (as part of the study)
Arm/Group | Gadobutrol (Gadavist, BAY 86-4875)
Serious Adverse Events (participants affected / at risk) | 1/479
Other Adverse Events (participants affected / at risk) | 0/479
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gadobutrol (Gadavist, BAY 86-4875) (N=479)
Cerebrovascular accident (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other